CLINICAL TRIAL: NCT00887432
Title: Randomized Placebo-Controlled, Double-Blind Study of Cholecalciferol Replacement in Patients on Expectant Management for Localized Prostate Cancer
Brief Title: Cholecalciferol Supplement in Treating Patients With Localized Prostate Cancer Undergoing Observation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: I 128308; NCI-2009-01530 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 128308 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH)
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Results first posted 2021-08-10 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Prostate Adenocarcinoma
MeSH Terms: interventions — Cholecalciferol; Watchful Waiting; Observation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (cholecalciferol and placebo) (Experimental): Patients receive cholecalciferol PO QD for 9 months in the absence of disease progression or unacceptable toxicity. After a wash-out period of 3 months, patients cross-over to Arm II.
  Interventions: Dietary Supplement: Cholecalciferol; Other: Laboratory Biomarker Analysis; Other: Patient Observation; Drug: Placebo Administration; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (placebo and cholecalciferol) (Experimental): Patients receive placebo PO QD for 9 months in the absence of disease progression or unacceptable toxicity. After a wash-out period of 3 months, patients cross-over to Arm I.
  Interventions: Dietary Supplement: Cholecalciferol; Other: Laboratory Biomarker Analysis; Other: Patient Observation; Drug: Placebo Administration; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Dietary Supplement: Cholecalciferol — Given PO
  Other Names: 9,10-Secocholesta-5,7,10(19)-trien-3-ol; Calciol; Delsterol; Vitamin D3
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Patient Observation
  Other Names: Active Surveillance; deferred therapy; expectant management; Observation; Watchful Waiting
Drug: Placebo Administration — Given PO
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized clinical trial studies how well cholecalciferol supplement works in treating patients with localized prostate cancer undergoing observation. Cholecalciferol may help prostate cancer cells become more like normal cells, and to grow and spread more slowly.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the prostate-specific antigen (PSA) response with oral high dose vitamin D3 supplementation (cholecalciferol) in patients with localized, histologically proven adenocarcinoma of the prostate who have not received any treatment for prostate cancer ever and have chosen expectant management.

SECONDARY OBJECTIVES:

I. To examine the pattern of response of PSA dynamics as well as the absolute change in PSA following vitamin D3 supplementation.

II. Assess the toxicity of vitamin D3 supplementation in men with prostate cancer.

TERTIARY OBJECTIVES:

I. Track occurrence of infections, deep venous thrombosis, vascular events and falls in the study population.

II. To evaluate relationship between cytochrome P450 family 24 (CYP24), 27B1, single-nucleotide polymorphism (SNPs) and serum 25(hydroxy [OH]) vitamin D response to oral D3 supplementation.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive cholecalciferol orally (PO) once daily (QD) for 9 months in the absence of disease progression or unacceptable toxicity. After a wash-out period of 3 months, patients cross-over to Arm II.

ARM II: Patients receive placebo PO QD for 9 months in the absence of disease progression or unacceptable toxicity. After a wash-out period of 3 months, patients cross-over to Arm I.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with clinically localized, histologically proven adenocarcinoma of prostate who has not received any treatment for prostate cancer ever and has chosen active surveillance; treatment for prostate cancer is defined as prostatectomy, androgen deprivation, brachytherapy or a full course of external beam irradiation
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Willingness to comply with study guidelines
* Willingness and ability to consent
* 25(OH) D3 level less than 40 ng/ml within 3 months of initiation of study; most recent 25 hydroxy D level within last 3 month would be used

Exclusion Criteria:

* History of malabsorption syndrome e.g., pancreatic insufficiency, celiac disease, tropical sprue
* Creatinine > 2.0 mg/dL
* Corrected serum calcium level of > 10.5 mg/dL (serum corrected calcium = serum calcium + 0.8[4-serum albumin])
* Most recent PSA value more than 18 months ago
* Prior or current therapy for prostate cancer
* Documented history of nephrolithiasis within the past 5 years
* Patients receiving finasteride (Proscar) or dutasteride (Avodart) or men who have received either agent within 90 days of entry are ineligible
* Patients cannot take any additional vitamin D supplementation during study treatment; patients taking > 2000 IU per day prior to treatment will be ineligible

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2009-04-08 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Mohler, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cholecalciferol to Placebo: Patients receive cholecalciferol PO QD for 9 months in the absence of disease progression or unacceptable toxicity. After a wash-out period of 3 months, patients cross-over to placebo PO QD for 9 months.
  Cholecalciferol: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Patient Observation
  Placebo Administration: Given PO
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
- Placebo to Cholecalciferol: Patients receive placebo PO QD for 9 months in the absence of disease progression or unacceptable toxicity. After a wash-out period of 3 months, patients cross-over to Cholecalciferol PO QD for 9 months.
  Cholecalciferol: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Patient Observation
  Placebo Administration: Given PO
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
Period: Overall Study
Arm/Group | Cholecalciferol to Placebo | Placebo to Cholecalciferol
Started | 58 | 74
Completed | 43 | 60
Not Completed | 15 | 14
Not completed — Start Excluded Therapy | 3 | 0
Not completed — Did not complete treatment | 6 | 8
Not completed — Protocol Violation | 2 | 3
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — No reason provided | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm I (Cholecalciferol and Placebo): Patients receive cholecalciferol PO QD for 9 months in the absence of disease progression or unacceptable toxicity. After a wash-out period of 3 months, patients cross-over to placebo PO QD for 9 months.
  Cholecalciferol: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Patient Observation
  Placebo Administration: Given PO
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
- Arm II (Placebo and Cholecalciferol): Patients receive placebo PO QD for 9 months in the absence of disease progression or unacceptable toxicity. After a wash-out period of 3 months, patients cross-over to cholecalciferol PO QD for 9 months.
  Cholecalciferol: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Patient Observation
  Placebo Administration: Given PO
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
- Total: Total of all reporting groups
Arm/Group | Arm I (Cholecalciferol and Placebo) | Arm II (Placebo and Cholecalciferol) | Total
Number analyzed (Participants) | 58 | 74 | 132
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 35 | 68
  >=65 years | 25 | 39 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (7.0) | 64.9 (6.5) | 64.3 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 58 | 74 | 132
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 50 | 69 | 119
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 58 | 74 | 132
Serum 25(OH)D3 [Mean (Standard Deviation); unit: ng/mL] — Baseline vitamin D measured in serum blood samples. Population: Lab values were not recorded for all patients.
  ng/mL
    number analyzed (Participants) | 18 | 21 | 39
    (all) | 25.1 (10.7) | 30.4 (9.0) | 27.9 (10.0)
Prostate Specific Antigen (PSA) [Mean (Standard Deviation); unit: ng/mL] — Population: The PSA at enrollment was not available for all subejcts.
  ng/mL
    number analyzed (Participants) | 57 | 72 | 129
    (all) | 5.2 (2.9) | 4.8 (2.6) | 5.0 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: PSA Response
Description: Difference in the mean change in PSA on vitamin D (9 month period: pre-Vitamin D to 9 months after start of vitamin D) versus on placebo (9 month period: pre-Placebo to 9 months after starting placebo).
  Compared using a paired t-test.
Time Frame: 9 month period: pre-Vitamin D/pre-placebo to 9 months after start of vitamin D/ placebo, up to 30 days after completion of study treatment
Population: Patients who completed both periods.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Cholecalciferol: Patients receive cholecalciferol PO QD for 9 months in the absence of disease progression or unacceptable toxicity.
  Cholecalciferol: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Patient Observation
  Placebo Administration: Given PO
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
- Placebo: Patients receive placebo PO QD for 9 months in the absence of disease progression or unacceptable toxicity.
  Cholecalciferol: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Patient Observation
  Placebo Administration: Given PO
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
Arm/Group | Cholecalciferol | Placebo
Number analyzed (Participants) | 87 | 87
ng/mL | 0.55 (2.13) | 0.31 (1.86)
Statistical Analysis 1: Comparison: Cholecalciferol vs Placebo; Evaluated the change in PSA under the vitamin D and placebo conditions using the combined data (n=87); Test type: Superiority; p = 0.431, t-test, 2 sided — Significance level of 0.05; Paired t-test, df=86; Mean Difference (Net) = 0.24, 95% CI 2-sided [-0.36 to 0.84]

2. Secondary Outcome: Slope of PSA Concentration Over Time
Description: The PSA levels were modeled as a function of treatment, time, their interaction, sequence, and a random subject effect using a linear mixed model. From this model, the subject specific PSA slope was obtained for each subject under each condition (vitamin D versus placebo). The PSA slopes were then compared between treatment conditions using linear mixed model to account for treatment arm and repeated measures.
Time Frame: 9 month period: pre-Vitamin D/pre-placebo to 9 months after start of vitamin D/ placebo, up to 30 days after completion of study treatment -Up to 30 days after completion of study treatment
Population: Including evaluable patients, those patients with data available under both the vitamin D and placebo conditions.
Measure: Least Squares Mean (Standard Error); unit: (ng/mL) / day
Arm/Group | Cholecalciferol | Placebo
Number analyzed (Participants) | 119 | 120
(ng/mL) / day | 0.000434 (0.000089) | 0.000245 (0.000090)
Statistical Analysis 1: Comparison: Cholecalciferol vs Placebo; Test type: Superiority — Comparing the mean PSA slopes between conditions (on vitamin D versus on placebo); p = 0.112, Mixed Models Analysis — Significance level of 0.05; Mean Difference (Net) = -0.00019, 95% CI 2-sided [-0.00042 to 0.000045]

3. Secondary Outcome: Toxicity as Assessed by National Cancer Institute Common Terminology Criteria for Adverse Events Version 3.0
Description: Summarizing the maximum observed treatment related adverse event. Summarize by arm and grade using frequencies and relative frequencies..
Time Frame: Up to 30 days after completion of study treatment (up to 22 months from start of study).
Population: All patients receiving any treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Cholecalciferol | Placebo
Number analyzed (Participants) | 119 | 120
Participants
  No AE | 117 | 118
  Grade 1 | 1 | 2
  Grade 2 | 0 | 0
  Grade 3 | 1 | 0
  Grade 4 | 0 | 0
  Grade 5 | 0 | 0

ADVERSE EVENTS:
Time Frame: Within 30 days of treatment completion (up to 22 months from start of study).
Arm/Group | Cholecalciferol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/119 | 0/120
Serious Adverse Events (participants affected / at risk) | 0/119 | 0/120
Other Adverse Events (participants affected / at risk) | 2/119 | 2/120
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cholecalciferol (N=119) | Placebo (N=120)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-26): https://cdn.clinicaltrials.gov/large-docs/32/NCT00887432/Prot_SAP_000.pdf